CLINICAL TRIAL: NCT03006588
Title: Fine Needle Aspiration of Retropharyngeal Lymph Node Guided by Endoscopic Ultrasound for the Diagnosis of Patients With Suspected Recurrent Nasopharyngeal Carcinoma
Brief Title: EUS-FNA for Retropharyngeal Lymph Node (RPLN) in Recurrent Nasopharyngeal Carcinoma (NPC) Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jian-jun Li, Associate Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EUS-FNA for RPLN(2016)
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: FNA,EUS,retropharyngeal lymph node (RPLN),NPC
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EUS-FNA for RPLN in NPC patients (Experimental): Fine needle aspiration guided by EUS in retropharyngeal lymph node in suspicious recurrent naspharyngeal carcinoma.
  Interventions: Procedure: EUS-FNA for RPLN in NPC patients

INTERVENTIONS:
Procedure: EUS-FNA for RPLN in NPC patients — An EUS probe was introduced to nasopharynx and the retropharyngeal space (RPS) were scanned. The suspicious recurrent RPLN, which was characterized as (1) roughly round and homogeneously hypo-echoic lesion in RPS; (2) located anterior to the carotid sheath which contained the internal carotid artery (ICA) and the internal jugular vein (IJV). Subsequently, guiding by EUS, a dedicated 22G needle was used to puncture into the enlarged RPLN, then the aspiration was conducted The entire EUS-FNA procedure was repeated at least three times till the satisfied strip tissue was obtained. The obtained tissue samples were sent for pathologic detection and the supernatant fluid was for thinprep cytologic test (TCT).

SUMMARY:
EUS-FNA for RPLN in NPC

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of a novel minimally invasive sampling technique -- fine needle aspiration (FNA) guided by endoscopic ultrasound (EUS), which aims to sample tissues from retropharyngeal lymph nodes (RPLN) for the diagnosis of patients with suspected recurrent nasopharyngeal carcinoma (NPC).

ELIGIBILITY:
Inclusion Criteria:

1. had undifferentiated, non-keratinizing carcinoma at the initial diagnosis (WHO, 1991 criteria) and no evidence of distant metastasis obtained before radiotherapy;
2. received regular chemotherapy with cytotoxic agents such as cisplatin, carboplatin, 5-fluorouracil, paclitaxel, etc, and coordinated with radiotherapy with standard doses (approximate 50-70 Gy) in nasopharynx and neck respectively. Within 3 months after radiotherapy, no local and distant lesions were found;
3. during regular follow-up , the enlarged RPLN was detected by MRI more than 6 months later since radiotherapy accomplished;
4. didn't receive chemotherapy radiotherapy, immunotherapy or salvage surgery from completion of radiotherapy to suspicious recurrent lesion in RPLN detected;
5. no recurrent lesion in nasopharynx was found by white light endoscopy as well as cancer cell negative in pathology by bite biopsy;
6. single lesion in RPLN, and no other recurrent or metastatic lesion was found in local region or distant organ.
7. the minimum axial diameter of RPLN was more than 5mm.

Exclusion Criteria:

* (1) patients with nasal stenosis; (2) patients with coagulation dysfunction; (3) patients with distant metastasis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy | Up to 24 weeks
  Number of participants with cancer positive and negative

CONTACTS AND LOCATIONS:
Overall Officials: Jian-jun Li, MD & Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No